CLINICAL TRIAL: NCT05927155
Title: Comparison of Bronchodilation and Oxygenation Patterns Induced by Long-acting β2-agonists and Muscarinic Antagonists in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of Acute Long-acting Bronchodilation on Oxygenation and Peripheral Ventilation in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Silvia Perez Bogerd, Chest physician, head of the COPD and Pulmonary Rehabilitation Clinic, Erasme University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SRB-201903-052; P2019/239 CCB: B406201939717 (Other: local ethics committee)
Record Dates: First submitted 2023-06-10; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting ß2-agonist; long-acting muscarinic antagonist; gas exchange; oxygen; small airways; lung capillary volume
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: A prospective, clinical, uncontrolled, single-blind, cross-over trial that included 2 visits over 2-3 days. Assessments were performed before and after long-acting bronchodilation (LABD): during the first visit, before, 30 minutes and 2 hours after inhalation of olodaterol (LABA); during the second visit, before, 40 minutes and 2 hours after the administration of 4 puffs of 2,5 µg of tiotropium (LAMA).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LABA (olodaterol) (Experimental): After 4-5 days washout period, during the first visit, participants received a long-acting beta2-agonist (LABA)
  Interventions: Drug: LABA
- LAMA (tiotropium) (Experimental): Two days after the first visit, during the second visit , participants received a long-acting muscarinic antagonist (LAMA)
  Interventions: Drug: LAMA

INTERVENTIONS:
Drug: LABA — Inhalation of 4 puffs of 2,5 µg of a long-acting beta2-agonist (LABA-olodaterol) administered via a spacer device
  Other Names: Olodaterol; Striverdi Respimat
  Arms: LABA (olodaterol)
Drug: LAMA — Inhalation of 4 puffs of 2,5 µg of a long-acting muscarinic antagonist (LAMA-tiotropium) administered via a spacer device
  Other Names: Tiotropium; Spiriva Respimat
  Arms: LAMA (tiotropium)

SUMMARY:
The goal of this clinical trial was to compare the action of long-acting ß2-agonists (LABA-olodaterol) and muscarinic antagonists (LAMA-tiotropium) on tissue oxygenation in COPD considering their impact on proximal and peripheral ventilation and, eventually, on lung capillary volume. The hypothesis was that LABA would have a more peripheral effect than LAMA (due to the opposite gradient of their receptors) and better peripheral ventilation would result in a greater oxygenation.

Before and after LABA (visit 1) and LAMA (visit 2) inhalation, COPD participants were asked to perform single-breath washout and forced oscillation tests, double diffusion technique and spirometry, while transcutaneous oxygenation was continuously recorded.

DETAILED DESCRIPTION:
Slopes of He (SHe) and SF6 (SSF6) from single-breath washout test (SBWO) (assessing ventilation heterogeneities at the level of pre- and intra-acinar bronchioles, respectively) (quadruple model, LR6000 Logan-Sinclair, Rochester, UK), respiratory system resistance (R5, R5-R19) and reactance (X5, AX, Fres) from forced oscillation test (FOT) (Resmon Pro, ResTech, Italy), lung capillary volume (Vc) from double diffusion of NO and CO (DLNO/DLCO) (Hyp'Air compact, Medisoft, Dinant, Belgium), and FEV1 from spirometry (Zan®, Oberthulba, Germany) were evaluated before and after LABD administered via a spacer device: during the first visit, before, 30 minutes and 2 hours after inhalation of 4 puffs of 2,5 µg of olodaterol (LABA); during the second visit, before, 40 minutes and 2 hours after the administration of 4 puffs of 2,5 µg of tiotropium (LAMA). Transcutaneous oximetry (Perimed232©, Järfälla, Sweden) was monitored continuously during the 2 hours of each visit.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to international criteria

Exclusion Criteria:

* inability to perform the tests or to maintain the washout period
* an exacerbation within the previous 6 weeks
* a diagnosis of asthma or another chronic respiratory disease that could influence the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation (TcO2) change from baseline | 120 minutes post-drug-administration
  Transcutaneous oxygen (TcO2) evaluated continuously with a transcutaneous oximeter
Tissue oxygenation (TcO2) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  Transcutaneous oxygen (TcO2) evaluated continuously with a transcutaneous oximeter

SECONDARY OUTCOMES:
Slope of Helium (SHe) change from baseline | 120 minutes post-drug administration
  SHe from single-breath washout test (SBWO) assessing peripheral ventilation heterogeneities
Slope of Helium (SHe) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  SHe from single-breath washout test (SBWO) assessing peripheral ventilation heterogeneities
Area under reactance curve from 5 Hz (AX) change from baseline | 120 minutes post-drug administration
  AX from forced oscillation test (FOT) evaluating the peripheral lung function
Area under reactance curve from 5 Hz (AX) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  AX from forced oscillation test (FOT) evaluating the peripheral lung function
Reactance at 5 Hz (X5) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  X5 from forced oscillation test (FOT) also evaluating the peripheral lung function
Resonant frequency (Fres) change from baseline | 120 minutes post-drug administration
  Fres from forced oscillation test (FOT) also evaluating the peripheral lung function
Resonant frequency (Fres) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  Fres from forced oscillation test (FOT) also evaluating the peripheral lung function
Peripheral resistance (R5-R19) change from baseline | 120 minutes post-drug administration
  Peripheral resistance, assessed as frequency dependence of resistance (R5-R19) from forced oscillation test (FOT) also evaluating the peripheral lung function
Peripheral resistance (R5-R19) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  Peripheral resistance, assessed as frequency dependence of resistance (R5-R19) from forced oscillation test (FOT) also evaluating the peripheral lung function
Lung capillary volume (Vc) change from baseline | 120 minutes post-drug administration
  Vc from single-breath double diffusion technique of nitric oxide (NO) and carbon monoxide (CO) (DLNO/DLCO)
Lung capillary volume (Vc) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  Vc from single-breath double diffusion technique of nitric oxide (NO) and carbon monoxide (CO) (DLNO/DLCO)
Forced Expiratory Volume in 1 Second (FEV1) change from baseline | 120 minutes post-drug administration
  FEV1 from spirometry
Forced Expiratory Volume in 1 Second (FEV1) change from baseline | 30 (LABA)/40 (LAMA) minutes post-drug administration
  FEV1 from spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Pérez Bogerd, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
When published, the datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the results
Access Criteria: The datasets used and/or analysed during the study will be available from the corresponding author on reasonable request.